CLINICAL TRIAL: NCT05709756
Title: Prevalence and Predictors of Esophageal Thermal Lesions in High-Power-Short-Duration Ablation of Atrial Fibrillation
Acronym: VISUAL-AF
Status: Completed | Type: Observational
Sponsor: Helios Health Institute GmbH (Other)
Responsible Party: Sponsor
Other Study IDs: 549/20-ek
Record Dates: First submitted 2023-01-24; First posted 2023-02-02 (Actual); Last update posted 2023-10-02 (Actual); Status verified 2023-01

CONDITIONS: Esophagus Injury; Atrial Fibrillation
Keywords: Atrial Fibrillation; Esophagus Injury; Pulmonary vein isolation; Esophagoscopy
MeSH Terms: conditions — Atrial Fibrillation

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Patients with documented atrial fibrillation who were referred to our clinic for catheter ablation will undergo standard HPSD ablation and subsequent esophagoscopy.

After esophagoscopy patients will be followed up for one month in the form of a telephone follow-up.

The primary endpoint of the study assessed by esophagoscopy performed on the day after the index catheter ablaton is the incidence of esophageal thermal lesions.

Secondary endpoints include:

1. The size of the esophageal thermal lesions.
2. The severity of esophageal thermal lesions.

ELIGIBILITY:
Inclusion Criteria:

* Atrial fibrillation documented in the 12-lead ECG
* Indication for catheter ablation in accordance with currentn ESC guidelines

Exclusion Criteria:

* Pregnancy
* Women of childbearing potential without a negative pregnancy test within 48 hours prior to ablation procedure
* Known intracardiac or other thrombi
* Contraindication to anticoagulation
* Contraindication to esophagoscopy: diseases and deformities of the cervical spine, esophageal varices

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients with documented atrial fibrillation who were referred to our clinic for pulomary vein isolation
Sampling Method: Non-Probability Sample
Enrollment: 263 (Actual)
Dates: Start 2021-03-01 (Actual); Primary Completion 2023-08-01 (Actual); Study Completion 2023-09-01 (Actual)

PRIMARY OUTCOMES:
Prevalence of ablation-related esophageal thermal lesions | One day after Catheter ablation
  It will be assessed by means of Esophagoscopy

SECONDARY OUTCOMES:
Size of ablation-related esophageal thermal lesions | One day after Catheter ablation
  It will be assessed by means of Esophagoscopy
Severity of ablation-related esophageal thermal lesions | One day after Catheter ablation
  It will be assessed by means of Esophagoscopy

CONTACTS AND LOCATIONS:
Overall Officials: Gerhard Hindricks, MD, Study Chair — Leipzig Heart Center at University of Leipzig; Arash Arya, MD, Study Director — Leipzig Heart Center at University of Leipzig
Locations (2):
- Germany (2):
  - Arash Arya, Leipzig, Saxony
  - Department of Electrophysiology, Leipzig Heart Center at University of Leipzig, Leipzig, Saxony

REFERENCES:
- [Derived] Wolff C, Langenhan K, Wolff M, Efimova E, Zachaus M, Darma A, Dinov B, Seewoster T, Nedios S, Bertagnolli L, Wolff J, Paetsch I, Jahnke C, Bollmann A, Hindricks G, Bode K, Halm U, Arya A. Incidence and predictors of thermal oesophageal and vagus nerve injuries in Ablation Index-guided high-power-short-duration ablation of atrial fibrillation: a prospective study. Europace. 2024 May 2;26(5):euae107. doi: 10.1093/europace/euae107. PMID 38646922